CLINICAL TRIAL: NCT05789121
Title: Effect of Rhythmic Auditory Stimulation (RAS) During Gait on Cortical Activation: A Functional Near-infrared Red Spectroscopy Neuroimaging Study (fNIRS)
Brief Title: Study of Cerebral Activation by fNIRS During Gait With Different Rhythmic Auditory Stimulations in Healthy Subjects
Acronym: MoveNIRS
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Other Study IDs: CHRO-2022-09
Record Dates: First submitted 2023-03-10; First posted 2023-03-29 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Healthy
Keywords: Rhythmic auditory stimulation; Gait; Near infrared spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy subjects: 30 healthy subject aged between 18 and 40.
  Interventions: Device: walking 25 m in 4 different conditions

INTERVENTIONS:
Device: walking 25 m in 4 different conditions — The protocol consisted of walking 25 m in 4 different conditions in the following order:
  Gait1, RAS-Slow, RAS-fast, Gait2.
  * Gait 1 : preferred cadence without auditory stimulation
  * RAS-Slow : Gait with low tempo rhythmic auditory stimulation by music (68.5 per minute).
  * RAS-Fast : Gait with fast tempo (10% above each Gait1 cadence).
  * Gait2 : preferred cadence without auditory stimulation

SUMMARY:
The purpose of this study is to investigate the cerebral activation in healthy subjects in 4 conditions of gait :

* Gait at preferred cadence without auditory stimulation (Gait1)
* Gait with low tempo rhythmic auditory stimulation by music (RAS-Slow). The beat rate of the music was 68.5 per minute for all participants.
* Gait with fast tempo synchronous rhythmic auditory stimulation by music (RAS-Fast). The beat rate of the music was set to 10% above each patient's preferred gait cadence . The preferred cadence was considered as the mean of the 6 trials during Gait 1.
* Gait without auditory stimulation (Gait2) The investigators goal is to compare cerebral activation and gait parameters during the 4 different tasks using fNIRS.

DETAILED DESCRIPTION:
Gait and balance impairments caused by neurological disorders affect many people around the world and impact on independent living and quality of life. Gait rehabilitation is therefore highly important for individuals with neurological diseases. In recent years, rehabilitation strategies were carried out considering new technological devices and paradigms have been developed to increase the effectiveness of rehabilitation. Brain and clinical research have provided a new understanding of the capabilities of music to engage and shape motor functions to support brain recovery processes. Humans possess an ability to perceive and synchronize movements to the beating music. In context of motor rehabilitation, musical rhythm entrains movement in patients with neurological impairment, opening new frontiers for using rhythm and music to prime the motor system and favour improvement of deficiency consequences. Rhythmic auditory stimulation (RAS) is a gait rehabilitation method in which patients synchronize foot steps to a metronome or musical beats. Typically, rhythmic cues are matched to the individual's preferred cadence and, once the movement is entrained to the external cues, the rhythm is gradually increased by 5-10% over baseline. However, little is known about the neural correlates of gait during RAS.

fNIRS (functional Near Infra Red Spectroscopy) is a functional method that allows to study the cerebral cortex changes during different tasks (like fMRI). This technique therefore makes it possible to study brain activation under more ecological conditions than fMRI and are therefore particularly suitable for exploring rehabilitation techniques.

This research aims to study and compare in healthy subjects, using, the brain regions involved in 4 conditions of gait without and with rhythmic auditory stimulations.

The protocol has 4 conditions :

* Gait at preferred cadence without auditory stimulation (Gait1)
* Gait with low tempo rhythmic auditory stimulation by music (RAS-Slow). The beat rate of the music was 68.5 per minute for all participants.
* Gait with fast tempo synchronous rhythmic auditory stimulation by music (RAS-Fast). The beat rate of the music was set to 10% above each patient's preferred gait cadence . The preferred cadence was considered as the mean of the 6 trials during Gait 1.
* Gait without auditory stimulation (Gait2) The investigators choosed a fixed order rather a randomized one, because the use of auditory stimulation may interferes with subsequent tasks. The comfortable gait was proposed as first and last conditions to check this aftereffect.

The fNIRS will used the Brite MKII apparatus. Gait parameters were recorded by FeetMe(R) Monitor (insole version FTM-DK, Atmel firmware version 2.3.10, Nordic firmware version 6.3.15).

Four gait parameters, including speed, cadence, stride length and double support time were analyzed. Gait speed is defined as the walking distance in a second (in cm/s), cadence as the number of steps within a minute walk (in steps/min). Stride length indicates the distance (in cm) from initial contact of one foot to subsequent contact of same foot. Double support time occurs when both feet are in contact with the ground simultaneously, it is normalized to stride time and expressed in % Gait Cycle (%). These 4 parameters are the most commonly used when studying the effect of SAR on gait.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 40 years old.
* No known neurological disease
* Benefiting from a social security coverage.
* Sufficient knowledge of the French language to understand the instructions

Exclusion Criteria:

* Person under tutorship or curatorship
* Known allergy to components of the fNIRS device: neoprene
* History of neurological disease
* History of rheumatological disease affecting walking
* Pregnant or breastfeeding women
* Subjects opposed to participating in the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy subjects aged between 18 and 40 years
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Mean change in the concentration of oxyhemoglobin during the task | Day 0
Mean change in the concentration of deoxyhemoglobin during the task | Day 0

SECONDARY OUTCOMES:
Walking speed | Day 0
Number of steps within a minute walk (in steps/min) | Day 0
  Number of steps within a minute walk (in steps/min)
stride length | Day 0
double support time | Day 0

CONTACTS AND LOCATIONS:
Overall Officials: Auzou PASCAL, Dr, Principal Investigator — CHR d'Orleans
Locations (1):
- CHR Orléans, Orléans, France

REFERENCES:
- [Background] Altenmuller E, Schlaug G. Apollo's gift: new aspects of neurologic music therapy. Prog Brain Res. 2015;217:237-52. doi: 10.1016/bs.pbr.2014.11.029. Epub 2015 Feb 11. PMID 25725918
- [Background] Bonnal J, Monnet F, Le BT, Pila O, Grosmaire AG, Ozsancak C, Duret C, Auzou P. Relation between Cortical Activation and Effort during Robot-Mediated Walking in Healthy People: A Functional Near-Infrared Spectroscopy Neuroimaging Study (fNIRS). Sensors (Basel). 2022 Jul 25;22(15):5542. doi: 10.3390/s22155542. PMID 35898041
- [Background] Braunlich K, Seger CA, Jentink KG, Buard I, Kluger BM, Thaut MH. Rhythmic auditory cues shape neural network recruitment in Parkinson's disease during repetitive motor behavior. Eur J Neurosci. 2019 Mar;49(6):849-858. doi: 10.1111/ejn.14227. Epub 2018 Dec 3. PMID 30375083
- [Background] Farid L, Jacobs D, Do Santos J, Simon O, Gracies JM, Hutin E. FeetMe(R) Monitor-connected insoles are a valid and reliable alternative for the evaluation of gait speed after stroke. Top Stroke Rehabil. 2021 Mar;28(2):127-134. doi: 10.1080/10749357.2020.1792717. Epub 2020 Jul 13. PMID 32654627
- [Background] Koshimori Y, Thaut MH. Future perspectives on neural mechanisms underlying rhythm and music based neurorehabilitation in Parkinson's disease. Ageing Res Rev. 2018 Nov;47:133-139. doi: 10.1016/j.arr.2018.07.001. Epub 2018 Jul 10. PMID 30005957
- [Background] Merchant H, Grahn J, Trainor L, Rohrmeier M, Fitch WT. Finding the beat: a neural perspective across humans and non-human primates. Philos Trans R Soc Lond B Biol Sci. 2015 Mar 19;370(1664):20140093. doi: 10.1098/rstb.2014.0093. PMID 25646516
- [Background] Thaut MH. The discovery of human auditory-motor entrainment and its role in the development of neurologic music therapy. Prog Brain Res. 2015;217:253-66. doi: 10.1016/bs.pbr.2014.11.030. Epub 2015 Feb 2. PMID 25725919